CLINICAL TRIAL: NCT06866171
Title: Phase II - Modular Convertible Child Safety Seat to Improve Usage
Brief Title: Swivel Convertible Child Safety Seat to Improve Usage
Status: Not yet recruiting | Type: Observational
Sponsor: Minnesota HealthSolutions (Industry)
Responsible Party: Principal Investigator, Julie Mansfield, Research Associate Professor, Minnesota HealthSolutions
Other Study IDs: MinnesotaHealthSolutions_Swiv
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Motor Vehicle Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study population: Participants must be a caregiver to a child age 4 or under, have experience installing a child safety seat within the past 2 years, and be physically healthy enough to install two child seats for the study.
  Interventions: Other: Modular child restraint

INTERVENTIONS:
Other: Modular child restraint — The participant will be asked to install two different child safety seats into a vehicle, presented to the participant one at a time (random order). The researcher will explain that the participant should install each seat to the best of his/her ability and may take as long as needed. When each installation is completed, the participant will be led away from the vehicle while their work is evaluated by a study-team approved researcher who is a certified Child Passenger Safety Technician (CPST). A data collection form will be used to document any installation errors. Following the installations, participants will complete a short survey with open-ended queries to describe facilitators or barriers they experienced while installing the seats, as well as what they liked or did not like about each seat. They will use a Likert scale to rate their self-efficacy in installing the seats, if they believed they were installed correctly, general ease-of-use, and which seat they preferred.

SUMMARY:
Child car safety seats (or "car seats") are an important tool to keep children safe in motor vehicle crashes, but are often misused by parents and caregivers. The installation of car seats can be time consuming and confusing. A new type of swivel car seat is being developed to potentially alleviate some of the typical frustrations that might lead to car seat misuse, specifically the visibility and usage of the top tether feature. This study aims to evaluate the new car seat product and determine whether the new design results in fewer installation errors compared to a traditional car seat.

Primary objective: To compare the number of top tether installation errors produced with a production-ready prototype swivel child safety seat vs. a traditional (control) seat.

Secondary objective: To assess self-reported preference and opinions on the swivel child safety seat design.

DETAILED DESCRIPTION:
Background: A preliminary Phase I study has already been conducted, in which volunteer focus groups provided qualitative feedback on a new prototype design. For this Phase II study, the revised prototype will be quantitatively and qualitatively evaluated by a larger sample of volunteers. Volunteer adult participants will be asked to complete two car seat installations: one with the new swivel prototype, and one with a traditional control car seat. Basic instruction manuals will be provided. The types and frequency of installation errors for each car seat will be quantified, and qualitative feedback on the product designs will be collected via survey.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65
* Care provider to a child who is up to 4 years of age
* Have installed a child safety seat in the last 2 years
* Able to lift and install a child safety seat into a vehicle
* English speaking.

Exclusion Criteria:

* Not meeting any of the above

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from the Central Ohio area. Adults who meet the above criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Correct use of top tether, prototype seat | 1 study visit, an average of 30 minutes
  Number of participants who correctly install the top tether in the prototype swivel seat
Correct use of top tether, traditional seat | 1 study visit, an average of 30 minutes
  Number of participants who correctly install the top tether in the traditional seat

SECONDARY OUTCOMES:
Correct overall installation, prototype seat | 1 study visit, an average of 30 minutes
  Number of participants who correctly install the prototype swivel child seat, considering all types of possible errors
Correct overall installation, traditional seat | 1 study visit, an average of 30 minutes
  Number of participants who correctly install the traditional child seat, considering all types of possible errors
Opinion on modular child seat design and instructions | 1 study visit, an average of 30 minutes
  Number of participants who rate the usability of the prototype swivel seat at least as high or higher than the traditional seat

CONTACTS AND LOCATIONS:
Overall Officials: Julie Mansfield, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be available upon request after publication of the results.